CLINICAL TRIAL: NCT07242040
Title: Sleep Disturbance and Daytime Fatigue as Predictors of Cognitive Decline and Functional Decline in Chronic Rhinosinusitis
Acronym: SNOOZE-CRS
Status: Completed | Type: Observational
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, lecturer, Sinai University
Other Study IDs: SU.REC.2025(58H)
Record Dates: First submitted 2025-09-26; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Rhinosinusitis; Sleep Disorders; Fatigue; Cognitive Dysfunction; Quality of Life Impairment
Keywords: Quality of Life; Functional Decline; Cognitive Decline; Daytime Fatigue; Sleep Disturbance; Chronic Rhinosinusitis
MeSH Terms: conditions — Sleep Wake Disorders; Fatigue; Cognitive Dysfunction; Parasomnias | interventions — Sleep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRS Patients Group: All participants were adults diagnosed with chronic rhinosinusitis (CRS). This group underwent standardized, non-interventional assessments to evaluate the association between sleep disturbance, daytime fatigue, and quality of life outcomes. No experimental treatment or diagnostic procedures were administered as part of the study.
  Interventions: Diagnostic Test: Self-Reported Questionnaires for Sleep, Fatigue, and Quality of Life

INTERVENTIONS:
Diagnostic Test: Self-Reported Questionnaires for Sleep, Fatigue, and Quality of Life — Participants completed a set of validated self-report instruments to assess:
  Sleep disturbance (Likert-type scale)
  Daytime fatigue (Likert-type scale)
  Quality of life - physical and mental domains
  No clinical intervention was introduced. Data were analyzed using correlation and regression models to determine predictive associations.

SUMMARY:
FOCUS-CRS is a cross-sectional observational study examining the relationship between sleep disturbance, daytime fatigue, and cognitive and functional health in patients with chronic rhinosinusitis (CRS). The study aims to determine whether self-reported sleep and fatigue scores predict impairments in physical and cognitive quality of life domains. A total of 134 adult CRS patients completed structured questionnaires assessing symptom burden and quality of life. Correlational and multivariate regression analyses were conducted to evaluate the predictive role of sleep disturbance and fatigue on functional and cognitive outcomes. This study seeks to improve understanding of underrecognized systemic effects of CRS, with implications for multidisciplinary patient care.

DETAILED DESCRIPTION:
Background:

Chronic rhinosinusitis (CRS) is a prevalent inflammatory condition associated with significant impairment in quality of life. While sinonasal symptoms are well-documented, systemic manifestations such as sleep disturbance, fatigue, and cognitive decline are underexplored. Emerging evidence suggests that sleep and energy dysregulation may independently contribute to cognitive dysfunction and physical debilitation in chronic inflammatory diseases. However, limited research has quantified these associations specifically in CRS.

Objective:

The FOCUS-CRS study (Fatigue and cOgnitive Comorbidities of chrOnic rSinosUS) investigates whether sleep disturbance and daytime fatigue are significant predictors of cognitive and functional decline in adults with CRS. The study also explores the role of demographic and clinical factors such as age, gender, duration of symptoms, and comorbid conditions in moderating these relationships.

Methods:

This is a single-center, cross-sectional observational study involving 134 CRS patients recruited from outpatient clinics. Participants completed validated questionnaires measuring sleep disturbance, daytime fatigue, and domain-specific quality of life (QoL), including physical functioning (QoL-physical) and cognitive/mental health (QoL-mental). Spearman correlations and multivariate linear regression were performed to assess the predictive effects of sleep and fatigue scores on QoL outcomes, controlling for potential confounders.

Expected Impact:

The findings from this study will enhance clinical awareness of sleep and fatigue-related comorbidities in CRS and support the development of integrative care models. Early identification and management of sleep and fatigue symptoms may contribute to improved cognitive and functional outcomes in CRS patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with CRS based on clinical guidelines
* Symptom duration ≥12 weeks
* Ability to provide informed consent

Exclusion Criteria:

* Prior sinus surgery
* Neurological or psychiatric disorders
* Use of sedatives or sleep-modulating medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study enrolled adult patients diagnosed with chronic rhinosinusitis (CRS), attending otolaryngology outpatient clinics at [insert institution name] during the study period. All participants met clinical diagnostic criteria for CRS as defined by current otolaryngologic guidelines (e.g., symptom duration ≥12 weeks, with or without radiologic confirmation). Eligible individuals were aged 18 years or older, capable of providing informed consent, and willing to complete standardized self-reported questionnaires related to sleep, fatigue, and quality of life. Patients with prior sinus surgery, neurological or psychiatric illness, or those on medications affecting sleep or cognition were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Quality of life scale | Day 1 (Single assessment at time of survey completion)
  The SF-36 Health Survey is a well-established instrument for measuring general health and quality of life. It evaluates eight domains of health, including both physical and mental aspects. Two summary scores are derived from these domains: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
  Physical Component Summary (PCS): Reflects physical health and functioning, including physical limitations and pain.
  Mental Component Summary (MCS): Reflects emotional well-being, social functioning, and mental health status.

SECONDARY OUTCOMES:
SNOT-22 Scale | Day 1 (Single assessment at time of survey completion)
  The SNOT-22 is a widely used instrument to evaluate the impact of sinonasal conditions (e.g., chronic rhinosinusitis) on quality of life. It consists of 22 questions that assess symptoms and how these symptoms interfere with daily activities. The questions cover aspects such as nasal symptoms, sleep disturbance, and the impact on social functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai university, Cairo, Egypt